CLINICAL TRIAL: NCT04124770
Title: Changes in Ultrasound-guided Skin Markings of the Cricothyroid Membrane in Three Different Neck Positions: a Prospective Observational Pilot Study
Brief Title: Neck Position and Ultrasound Landmark of Cricothyroid Membrane
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christopher Prabhakar, Clinical Assistant Professor, University of British Columbia, University of British Columbia
Other Study IDs: H18-01601
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Cricothyroid Membrane; Ultrasound; Airway; Cricothyroidotomy
MeSH Terms: interventions — Movement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Movement — Re-positioning of neck

SUMMARY:
Cricothyroid membrane (CTM) localization is a critical step prior to emergent surgical airway access. Ultrasound-guided localization of the CTM on the skin of the neck had been suggested prior to induction of general anesthesia so that a marked entry point can be used to quickly establish emergent front of neck access if required. In this prospective observational study, the investigators aim to determine the potential for migration of the CTM markings in the sagittal plane during neck repositioning.

DETAILED DESCRIPTION:
As defined in recent difficult airway guidelines, successful and rapid cricothyroidotomy depends on identification of the cricothyroid membrane (CTM), coupled with skillful and efficient technique. Unfortunately, identification of the CTM is often inaccurate and complicated by patient factors such as female gender and obesity. Further studies go on to demonstrate the rates for correct identification of the CTM using palpation methods are low and range between 11% and 42%, with even lower success of identifying the midline of the CTM. This traditional palpation method was demonstrated to be fraught with error by different users including: 2 finger palpation, 4 finger palpation, and neck crease successfully identified the CTM 62%, 46%, and 50% of the time at time intervals between 11-14 seconds in non emergency settings.

As a result of previously mentioned patient factors and multiple technical factors, including poor landmarking, cricothyrotomy has a failure rate as high as 60%, exposing patients to high risks of mortality and morbidity. Therefore, more accurate methods of CTM identification are greatly needed at present.

Suggestions of implementing ultrasound in airway management have been brought forth, with applications such as predicting airway difficulty prior to instrumentation, confirming endotracheal tube position, or marking the CTM prior to induction of anesthesia. There have been multiple studies addressing questions such as mean time to identification of CTM in obese subjects using ultrasound and comparison of transverse versus longitudinal scanning technique. One group assessed translational movement of the CTM in neutral neck position versus extended in 23 healthy volunteers, and found a difference in transverse and longitudinal markings of 0.91mm and 1.04mm respectively, with CTM length ranging from 10.6mm to 17mm.

Of interest to the investigators is using ultrasound to predict CTM position accurately and ensuring ability to gain emergency airway access, as the accuracy of ultrasound identification of the CTM in different neck positions is unknown. What is specifically unknown is the translational movement of the cricoid between neck positions.

Therefore, the investigators propose an observational prospective trial looking at cricoid cartilage translation with three different neck positions: neck neutral, neck extension, and neck sniffing. The investigators will use GE Venue 50 (GE HealthcareTM) ultrasound machine, and a linear transducer probe with a frequency of 8-13MHz (GE LOGIQ 12L-SC) for measurements. The measurements will originate at the sternal notch to the superior border of the cricoid cartilage where the cricoid membrane inserts. These will also be referenced to exterior skin markings. The outcomes will address if the airway significantly moves during manipulation by the degree of cricoid cartilage translation between neutral, sniffing and extended neck positions. Secondarily, The investigators will also aim to address the directionality of a pre-marked neck and cricoid migration with neck manipulation.

ELIGIBILITY:
Inclusion

* Patients aged between 19 and 90
* Scheduled for elective surgeries

Exclusion

* history of cricothyrotomy
* history of tracheostomy
* history of thyroidectomy
* history of plastic surgery or neck skin flaps
* history of neck lymph node dissections
* history of open carotid endarterectomy
* history of cervical instrumentation
* history of neck deformities (acquired or congenital)
* history of allergic reactions to adhesive tapes.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult volunteers over age 19
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

PRIMARY OUTCOMES:
Cricothyroid membrane movement measured with ultrasound | 14 months
  The primary outcome was the distance measured from superior border of the cricoid cartilage to the sternal notch in the sagittal plane between the three neck positions

SECONDARY OUTCOMES:
Directionality of cricothyroid membrane movement measured by ultrasound | 14 months
  Directionality of the movement of the CTM during neck positions in relation to the sternal notch

CONTACTS AND LOCATIONS:
Locations (1):
- St Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participants data.

REFERENCES:
- [Background] Frerk C, Mitchell VS, McNarry AF, Mendonca C, Bhagrath R, Patel A, O'Sullivan EP, Woodall NM, Ahmad I; Difficult Airway Society intubation guidelines working group. Difficult Airway Society 2015 guidelines for management of unanticipated difficult intubation in adults. Br J Anaesth. 2015 Dec;115(6):827-48. doi: 10.1093/bja/aev371. Epub 2015 Nov 10. PMID 26556848
- [Background] Law JA, Broemling N, Cooper RM, Drolet P, Duggan LV, Griesdale DE, Hung OR, Jones PM, Kovacs G, Massey S, Morris IR, Mullen T, Murphy MF, Preston R, Naik VN, Scott J, Stacey S, Turkstra TP, Wong DT; Canadian Airway Focus Group. The difficult airway with recommendations for management--part 2--the anticipated difficult airway. Can J Anaesth. 2013 Nov;60(11):1119-38. doi: 10.1007/s12630-013-0020-x. Epub 2013 Oct 17. PMID 24132408
- [Background] Aslani A, Ng SC, Hurley M, McCarthy KF, McNicholas M, McCaul CL. Accuracy of identification of the cricothyroid membrane in female subjects using palpation: an observational study. Anesth Analg. 2012 May;114(5):987-92. doi: 10.1213/ANE.0b013e31824970ba. Epub 2012 Feb 24. PMID 22366848
- [Background] Lamb A, Zhang J, Hung O, et al. Exactitude du repérage de la membrane cricothyroïdienne par des stagiaires et des patrons en anesthésie dans un établissement canadien. Can J Anesth. 2015. doi:10.1007/s12630-015-0326-y.
- [Background] Katz JA. 4th National Audit Project of the Royal College of Anaesthetists and The Difficult Airway Society. Anesthesiology. 2012. doi:10.1097/ALN.0b013e31823cf122.
- [Background] Elliott DS, Baker PA, Scott MR, Birch CW, Thompson JM. Accuracy of surface landmark identification for cannula cricothyroidotomy. Anaesthesia. 2010 Sep;65(9):889-94. doi: 10.1111/j.1365-2044.2010.06425.x. PMID 20645953
- [Background] Bair AE, Chima R. The inaccuracy of using landmark techniques for cricothyroid membrane identification: a comparison of three techniques. Acad Emerg Med. 2015 Aug;22(8):908-14. doi: 10.1111/acem.12732. Epub 2015 Jul 21. PMID 26198864
- [Background] Cook TM, Woodall N, Frerk C; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 1: anaesthesia. Br J Anaesth. 2011 May;106(5):617-31. doi: 10.1093/bja/aer058. Epub 2011 Mar 29. PMID 21447488
- [Background] Kristensen MS, Teoh WH, Rudolph SS, Hesselfeldt R, Borglum J, Tvede MF. A randomised cross-over comparison of the transverse and longitudinal techniques for ultrasound-guided identification of the cricothyroid membrane in morbidly obese subjects. Anaesthesia. 2016 Jun;71(6):675-83. doi: 10.1111/anae.13465. Epub 2016 Apr 2. PMID 27037981
- [Background] Mallin M, Curtis K, Dawson M, Ockerse P, Ahern M. Accuracy of ultrasound-guided marking of the cricothyroid membrane before simulated failed intubation. Am J Emerg Med. 2014 Jan;32(1):61-3. doi: 10.1016/j.ajem.2013.07.004. PMID 24475485